CLINICAL TRIAL: NCT05599555
Title: Community-based Sero-epidemiological Study of COVID-19 to Provide Data in Real Time on Age-stratified Infection Attack Rates, Disease Severity and Population Immunity, for Guiding Intervention Policy
Brief Title: Community-based Sero-epidemiological Study of COVID-19
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 20-132
Record Dates: First submitted 2022-10-28; First posted 2022-10-31 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood donor serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unvaccinated blood donors: Blood donors who were unvaccinated with any COVID-19 vaccine by study recruitment
- Blood donors vaccinated with BNT162b2: Blood donors who were vaccinated with one or more doses of the mRNA vaccine Comirnaty (BNT162b2 mRNA, BioNTech/Fosun-Pharma, Mainz, Germany/Shanghai, China) by study recruitment.
  Interventions: Biological: mRNA BNT162b2 vaccine
- Blood donors vaccinated with CoronaVac: Blood donors who were vaccinated with one or more doses of the inactivated CoronaVac (Sinovac life Sciences, Beijing, China) vaccine by study recruitment.
  Interventions: Biological: CoronaVac vaccine

INTERVENTIONS:
Biological: mRNA BNT162b2 vaccine — mRNA vaccine Comirnaty (BNT162b2 mRNA, BioNTech/Fosun-Pharma, Mainz, Germany/Shanghai, China)
  Groups: Blood donors vaccinated with BNT162b2
Biological: CoronaVac vaccine — Inactivated CoronaVac vaccine (Sinovac Life Sciences, Beijing, China)
  Groups: Blood donors vaccinated with CoronaVac

SUMMARY:
Using detailed serial cross-sectional estimates of the age-specific distribution of SARS-CoV-2 Omicron variant-specific antibody positivity levels, the investigators derived age-specific infection attack rates and age-specific population immunity levels and tracked the magnitude of individual-level and population-level waning immunity over time. The findings will inform health policy makers on devising future public health and social measures and vaccination guidance in response to the ongoing COVID-19 pandemic.

DETAILED DESCRIPTION:
Since December 2021, the SARS-CoV-2 B.1.1.529 (Omicron) variant started spreading in Hong Kong, leading to an unprecedented 5th wave. It is known that the Omicron variant may partially evade immunity from past vaccination and infection although both appear to protect from severe disease and death. As Hong Kong emerges from the 5th wave, it will be critically important for public health policy to assess the proportion of the population with evidence of natural infection and those with evidence of detectable neutralizing antibody to the Omicron variant, either though natural infection or vaccination. Our project aims to assess these parameters.

The investigators recruited healthy blood donors by convenience sampling at the five largest blood donation centres (Mongkok, Causeway, Kwun Tong, Tsuen Wan and Shatin) of the Hong Kong Red Cross Blood Transfusion Service (HKRCBTS). Blood donors were matched by the HKRCBTS and the Hong Kong Department of Health with official vaccination records via unique Blood Transfusion Service donor identification numbers. The records were then anonymised and provided to the study team. Blood donors were also provided with the option of self-reporting their vaccination and COVID-19 infection history.

Since the investigators need to distinguish past infection from vaccine induced immunity, they used serological test strategies that would differentiate natural infection from vaccine immunity. The investigators have previously shown that IgG antibody to the Nucleocapsid protein of SARS-CoV-2 (whole protein and the C-terminal domain) provides evidence of past infection and is not elicited by BNT162b2 vaccine but may be elicited by CoronaVac vaccine (Wu et al. 2021, Mok et al. 2021) . They have also shown IgG antibody to ORF8 is elicited by past infection and not by either CoronaVac or BNT162b2 (Hachim et al. 2020). The investigators used these assays to assess evidence of natural infection in blood donor samples.

Through the above procedures, the investigators obtained detailed serial cross-sectional (weekly between mid-April and the end of July, followed by monthly until the end of 2022) estimates of the age-specific distribution of SARS-CoV-2 Omicron variant-specific antibody positivity levels. The investigators derived age-specific infection attack rates and age-specific population immunity levels and tracked the magnitude of individual-level and population-level waning immunity over time.

ELIGIBILITY:
Eligibility criteria follows criteria for blood donation in Hong Kong:

Inclusion Criteria:

* Have good health
* Weigh 41 kg or above (90 lbs or above)
* Aged between 18 and 65

Exclusion Criteria:

- Individuals who are not eligible for blood donation in Hong Kong

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy blood donors in Hong Kong aged between 18 and 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 9600 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Covid-19 seropositivity | 28 April 2022 to 31 December 2022
  Study subject is seropositive with SARS-CoV-2 anti-N (unvaccinated or BNT162b2 vaccinated donors only) or anti-ORF8 (CoronaVac vaccinated donors only) antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Wu, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No